CLINICAL TRIAL: NCT00919295
Title: Study of Anti-nociceptive Biogenic Amine Status, Indoleamine 2,3-dioxygenase Activity, Serum Levels of Cytokines, BDNF, BH4 and Mirtazapine Efficacy in Thai Fibromyalgia Syndrome Patients.
Brief Title: Study of Indoleamine 2,3-dioxygenase Activity, Serum Levels of Cytokines, BDNF, BH4 and Mirtazapine Efficacy in Fibromyalgia Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: University of Texas (Other); University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Suwimon Yeephu, Faculty of Pharmacy, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 323/2551(EC4)
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia syndrome; mirtazapine; randomized controlled trial; pilot study
MeSH Terms: conditions — Fibromyalgia | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo
- mirtazapine 15 (Placebo Comparator): mirtazapine 15 mg
  Interventions: Drug: mirtazapine
- mirtazapine 30 (Placebo Comparator): mirtazapine 30mg
  Interventions: Drug: mirtazapine

INTERVENTIONS:
Drug: mirtazapine — mirtazapine 15 mg or 30 mg tablet daily at bedtime for 13 weeks
  Other Names: Remeron
  Arms: mirtazapine 15; mirtazapine 30
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This study aims to investigate the anti-nociceptive biogenic amine (serotonin [5-hydroxytryptamine; 5-HT], norepinephrine [NE], dopamine [DA], and their metabolites) status, and serum levels of cytokines, BDNF and BH4 in Thai fibromyalgia syndrome (FMS) patients compared with a representative Thai population. The efficacy and the tolerability of mirtazapine as monotherapy for FMS will also be assessed. In addition, proof of concept of the indoleamine 2,3-dioxygenase (IDO) activity in FMS will be conducted.

The study will be divided into three parts. In part I, FMS patients of Thai ethnicity will be examined to determine the blood and/or urinary level of anti-nociceptive biogenic amines, cytokines, BDNF and BH4 by comparison with the demographically matched, but unrelated, healthy normal controls (HNC). In part II, the FMS subjects from part I study will be randomized to blinded therapy with mirtazapine or identical appearing placebo. There will be three treatment groups (N=1:1:1) to accommodate two dosages of mirtazapine (15 mg, 30mg) and placebo given before bedtime. Pill counts at baseline and at follow-up visits will document compliance. Standard outcome instruments (translated and validated in Thai language) will be used at baseline and at each of the follow-up visits. The co-primary outcome variable will be the changes in the pain visual analog scale (PVAS) score and pain responders (>= 30% PVAS reduction). Secondary clinical outcome variables of interest will include depression, insomnia, anxiety, physical function, morning stiffness, patient global assessment of disease status, patient global impression of change, fibromyalgia impact questionnaire (FIQ, quality of life and adverse experience. The changes of biogenic amine and IGF-1 concentrations in blood and/or urine with the treatment will be examined as the secondary biochemical measures. In part III, the IDO activity of depressed FMS, non-depressed FMS and HNC will be compared. Moreover, the effect of mirtazapine treatment on the IDO activity in depressed and non-depressed FMS patients will be assessed.

Study hypothesis

1. Anti-nociceptive biogenic amine levels in Thai FMS patients are lower than in Thai healthy normal control.
2. Higher IDO activity could be observed in FMS patients.
3. Higher cytokines could be observed in FMS patients.
4. Higher BDNF could be observed in FMS patients.
5. Lower BH4 could be observed in FMS patients.
6. Mirtazapine is effective in FMS treatment.

ELIGIBILITY:
Inclusion Criteria for randomized controlled trial:

* male or female outpatients > 18 years of age, descended from Thai parents
* meet criteria for FMS as defined by the American College of Rheumatology 1990
* have a score of > 4 on the pain visual analog scale (PVAS) score at screening

Exclusion Criteria:

* any severe or unstable physical or psychiatric disorder
* inflammation or injury or trauma in the previous month
* substance abuse within the past year
* serious suicide risk
* pregnancy or breastfeeding
* subject has an allergic reactions to mirtazapine or any of its constituents or severe allergic reactions to multiple medications
* comorbid inflammatory rheumatic diseases
* Use of medications or herbal agents with CNS activity
* regular use of analgesics with the exception of acetaminophen up to 2 gram/day
* chronic use of sedatives/hypnotics
* unable to discontinue medications that may affect the study results (all antidepressants, mood stabilizers, antipsychotics, sleep aids such as hypnotics, tranquilizers, sedating antihistamine and benzodiazepines, all analgesics including anticonvulsants, muscle relaxants, stimulant medications such as dextroamphetamine and methylphenidate, any other medications taken by the subject for the treatment of fibromyalgia
* unable to attend the follow-up schedule of the study
* not agree with avoidance or stable maintenance of unconventionalor alternative therapies, such as Thai traditional massage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-12; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for part II of this study will be "change from baseline in the severity of the pain visual analog scale (PVAS) score" and pain responders (>= 30% PVAS reduction). | day 7, 21, 35, 63, 91 (day 0 = first day of starting expected dose)

SECONDARY OUTCOMES:
Depression, sleep quality, patient global assessment of disease status, FIQ, PGIC, quality of life, adverse events | day 7, 21, 35, 63, 91 (day 0 = the day of starting expected dose)

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Yeephu, Principal Investigator — Faculty of Pharmacy Mahidol University; Saithip Suttiruksa, Master, Principal Investigator — Faculty of Pharmacy, Mahidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand